CLINICAL TRIAL: NCT02574559
Title: Cognitively Based Compassion Training for Parents of Children With Autism Spectrum Disorders
Brief Title: CBCT for Parents of Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel Fernandez-Carriba, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00074454
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Stress
Keywords: Caregiver; Stress; Depression; Autism Spectrum Disorder; Compassion Meditation
MeSH Terms: conditions — Depression; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caregiver of Child With Autism Spectrum Disorder (Experimental): Caregivers attending eight weekly sessions of Cognitive Based Compassion Training Sessions and Meditation.
  Interventions: Behavioral: Cognitive Based Compassion Training Session: Developing Attention and Stability of Mind; Behavioral: Cognitive Based Compassion Training Session: Cultivating Insight into the Nature of Mental Experience; Behavioral: Cognitive Based Compassion Training Session: Self-compassion; Behavioral: Cognitive Based Compassion Training Session: Cultivating Equanimity; Behavioral: Cognitive Based Compassion Training Session: Developing Appreciation and Gratitude for Others; Behavioral: Cognitive Based Compassion Training Session: Developing Affection and Empathy; Behavioral: Cognitive Based Compassion Training Session: Realizing Wishing and Aspiring Compassion; Behavioral: Cognitive Based Compassion Training Session: Realizing Active Compassion; Behavioral: Meditation Session

INTERVENTIONS:
Behavioral: Cognitive Based Compassion Training Session: Developing Attention and Stability of Mind — Completed at Week 1. Initial meditation exercises will be described and practiced to train attention skills (on breath) and create mental stability.
Behavioral: Cognitive Based Compassion Training Session: Cultivating Insight into the Nature of Mental Experience — Completed at Week 2. Exercises to develop mindfulness will continue in order to promote mental stability and clarity.
Behavioral: Cognitive Based Compassion Training Session: Self-compassion — Completed at Week 3: Techniques to analyze mental processes are introduced.
Behavioral: Cognitive Based Compassion Training Session: Cultivating Equanimity — Completed at Week 4. Further analysis of mental processes.
Behavioral: Cognitive Based Compassion Training Session: Developing Appreciation and Gratitude for Others — Completed at Week 5. A reflection of all the things that bring us well-being are provided by or dependent upon other beings is encouraged.
Behavioral: Cognitive Based Compassion Training Session: Developing Affection and Empathy — Completed at Week 6. The following concepts are presented and carefully considered: (1) cooperation and solidarity is essential for our survival and flourishing, as we are all extremely vulnerable and need each other; (2) hate and selfishness only cause suffering to others and ourselves and can only be prevented by cultivating sincere affection for others.
Behavioral: Cognitive Based Compassion Training Session: Realizing Wishing and Aspiring Compassion — Completed at Week 7. Participants are invited to deepen their reflection on the reasons for gratitude, empathy, and affection for others, and see how they lead to feelings of compassion, or the wish for others to be free from suffering.
Behavioral: Cognitive Based Compassion Training Session: Realizing Active Compassion — Completed at Week 8. The strategies used until this point will be reviewed in order to move from the wish for others to be free of suffering, toward the sense that we want to and must take steps to relieve their suffering.
Behavioral: Meditation Session — 20 minute session completed weekly after the Cognitive Training Session

SUMMARY:
The purpose of this study is to determine if caregivers of children with a developmental delay experience a decrease in stress by participating in a meditation/cognitive training protocol.

DETAILED DESCRIPTION:
A pilot-test, eight week, Cognitive Based Compassion Training (CBCT) program for caregivers of children with developmental delays that is comprised of eight two-hour weekly long sessions with a certified instructor followed by a twenty minute long meditation session. Sessions will focus on developing attention and stability of mind through focused attention training; cultivating insight into the nature of mental experience; cultivating self-compassion; developing equanimity; developing appreciation and gratitude; developing affection and empathy; realizing aspirational compassion; and realizing active compassion.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of child(ren) with developmental delay (including parents, grandparents, other extended family, family friends, and providers)
* Spend significant amount of time (more than 10 hours/week) with children with special needs.

Exclusion Criteria:

* Started to use any psychotropic medication within one year.
* Had any changes in any psychotropic medication doses taken within one year.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02-11 (Actual); Study Completion 2016-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  Designed to assess behavior problems in children with developmental difficulties and it consists of 58 items grouped in five subscales (irritability, social withdrawal, stereotypic behaviors, hyperactivity, and inappropriate behavior). The irritability subscale comprises of 15 statements that have been used as an index of Autism Spectrum Disorder-specific disability.

SECONDARY OUTCOMES:
Change in Parenting Stress Index/Short Form (PSI/SF) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A 36-item measure designed to evaluate the magnitude of stress in caregiver-child relationships. All items have a 5-point response scale (roughly, Strongly Agree, Agree, Not Sure, Disagree, Strongly Disagree) and yield a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child.
Change in Perceived Stress Scale (PSS) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  An instrument to measure non-specific appraised stress which correlates with biological markers like cortisol, immune markers, and depression. It consists of 14 items rated on a 5 point scale (from never to very often) that refer to feelings and thoughts over the past month.
Change in Acceptance and Action Questionnaire (AAQ) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A list of 10 statements rated from 1 (never true) to 7 (always true) measures psychological acceptance or assent to the reality of a situation (e.g., "it's okay if I remember something unpleasant").
Change in Interpersonal Reactivity Index (IRI) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A self-report questionnaire of 28 items answered on a 5-point scale ranging from "Does not describe me well" to "Describes me very well". It is considered a measure of empathy as a multidimensional construct that can be factored in four first-order factors, corresponding to the four subscales of the IRI: Perspective Taking, Fantasy (or tendency to transpose into the feelings and actions of fictitious characters in books and movies), Empathic Concern (interpersonal sympathy and concern), and Personal Distress (interpersonal distress).
Change in Mindful Attention Awareness Scale (MAAS) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A questionnaire to measure attentiveness and mindfulness as a trait and it includes 15 items with answers on a 6-point scale (from "almost always" to "almost never").
Change in Behavior Rating Inventory of Executive Function- Adult Version (BRIEF-A) Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A self-report assessment of executive function behaviors for adults aged 18-90. It contains 86 items in two validity scales and eight clinical scales that form two indexes: a) Behavioral Regulation (four scales: inhibit, shift, emotional control, and self-monitor) and b) Metacognition (five scales: initiate, working memory, plan/organize, organization of materials, and monitor), as well as a Global Executive Composite score.
Change in Parenting Sense of Competence Scale Score | Baseline, Completion of Treatment (up to eight weeks), Follow-Up (up to three months post-participation)
  A 16 item questionnaire (on a 6 point scale ranging from strongly agree to strongly disagree), it includes a section on Satisfaction, with nine questions that examine the parents' anxiety, motivation and frustration, and an Efficacy scale, with 7 questions covering parents' sense of competence, capability levels, and problem-solving abilities in their parenting role.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Fernandez-Carriba, PhD, Principal Investigator — Emory University Assistant Professor
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia